CLINICAL TRIAL: NCT00846664
Title: Increase in Multifidus Size By Short Arc Banding on the ATM Machine as Measure by Diagnostic Ultrasound
Brief Title: Short Arc Multifidus Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. Adam Morrell, Logan College of Chiropractic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR0112080162; 396
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Multifidus Disuse Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): Group 1 wil perform short arc banding twice a week for four weeks and have diagnostic ultrasound of multifidus measured before and after intervention
  Interventions: Procedure: Logan Short Arc Banding

INTERVENTIONS:
Procedure: Logan Short Arc Banding — Group 1 wil perform short arc banding twice a week for four weeks and have diagnostic ultrasound of multifidus measured before and after intervention

SUMMARY:
Patients will be performing Logan short arc banding protocols to see the effect on multifidus size

DETAILED DESCRIPTION:
The subjects will initially be scanned by diagnostic ultrasound by to assess the cross sectional area of their lumbar multifidi. Then they will perform 3 sets of 30 second periods of Logan Short Arc Banding on the ATM machine twice a week for 4 weeks and then they will be scanned again using diagnostic ultrasound to assess the effects of the rehabilitation exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ages 18-54

Exclusion Criteria:

* Asymptomatic of: Low Back Pain, previous spinal injury, surgery or other condition affecting the spine, local infection, injury or malignancy; pregnancy or any condition affecting muscle reaction time.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Multifidus cross sectional area | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States